CLINICAL TRIAL: NCT05403073
Title: Ultrasound Guided Nerve Block for Hip Fracture Pain Management at Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Borja Alcobía-Díaz MD, PhD, MD, PhD, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/027-EC_X
Record Dates: First submitted 2022-02-25; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Hip Fractures; Pain, Acute; Ultrasound Therapy; Complications
Keywords: Hip Fractures Pain Ultrasound nerve block
MeSH Terms: conditions — Hip Fractures; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Nerve Blocking (No Intervention): Pain management at ER Department will be as usually with iv drugs and 3 kilogram soft traction.
- Ultrasound Nerve blocking (Active Comparator): Pain management at ER Department will be as usually with iv drugs and ultrasound guided Suprainguinal Iliac Fascia Nerve Block.
  Interventions: Procedure: Ultrasound guided Suprainguinal Iliac Fascia Nerve Block.

INTERVENTIONS:
Procedure: Ultrasound guided Suprainguinal Iliac Fascia Nerve Block. — Pain management at ER Department will be as usually with iv drugs and ultrasound guided Suprainguinal Iliac Fascia Nerve Block.
  Arms: Ultrasound Nerve blocking

SUMMARY:
The main objective is to determine if ultrasound guided suprainguinal iliac fascia block leads in better clinical outcomes such as pain management or time to home discharge.

DETAILED DESCRIPTION:
Determining effectiveness in ultrasound guided suprainguinal iliac fascia block as a tool of comfortability of patients with less use of opioids and their side effects and its possible influence in early discharge to home has no evidence in orthopedics literature till today.

Ultrasound becomes an accessible tool at Emergency Departments and Orthopedic Surgeons are increasingly interested its clinical use.

This clinical trial wants to investigate if its use for hip nerve block leads in better clinical outcomes such as pain management or time to home discharge.

ELIGIBILITY:
Inclusion Criteria:

* Low energy Hip Fracture

Exclusion Criteria:

* Don´t meet Inclusion Criteria
* Present any other synchronic fracture.
* Drug allergy for drugs used for nerve blocking
* Skin infection at injection site.
* Contraindication due to comorbidities.
* Pathologic fractures.
* Cognitive impairment
* Do not give his consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Pain Control after Ultrasound guided nerve block vs iv painkillers | During Emergency Department stay (up to 12 hours)
  Using Visual Analogue Scale (1-No pain; 10 -worst pain) measure difference between pain during arrival at Emergency Department and 30 minutes after Ultrasound guided nerve block vs iv painkillers

SECONDARY OUTCOMES:
Patient Hip Mobility with tolerable pain | Immediately Before Discharging home assessed up to 2 weeks.
  Range of Motion Degrees
Functionality: Sit to Stand Test | Immediately Before Discharging home assessed up to 2 weeks.
  The 30-second chair stand involves recording the number of stands a person can complete in 30 seconds
Opioid Use | Immediately Before Discharging home assessed up to 2 weeks.
  Quantity of Opioid drugs consumed during Hospital stay expressed in Morphine equivalent doses
Patient Satisfaction | Immediately Before Discharging home assessed up to 2 weeks.
  Patient subjective satisfaction in a numeric scale from 1 (completely dissatisfied with pain management) to 10 (highest possible satisfaction with pain management).

CONTACTS AND LOCATIONS:
Overall Officials: Borja Alcobía-Díaz, MD, PhD, Principal Investigator — Clinical Assistant

IPD SHARING:
Plan to Share IPD: No
Email Contact